CLINICAL TRIAL: NCT05870072
Title: The Effect of Kinesthetic Motor Imagery Training and Dual Task Training on Cognitive and Motor Functions in Healthy Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevtap Cakir, Principal Investigator, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSBU-SEVTAP-0001
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Imagery, Psychotherapy; Exercise; Stroop Test; Healthy Participants; Multi-Tasking Behavior; Balance, Postural; Motor Activity; Cognitive Function; Cognitive Rehabilitation; Cognitive Test
MeSH Terms: conditions — Motor Activity; Multitasking Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual task training (balance exercises combined with cognitive task) group (Experimental)
  Interventions: Other: Dual task training
- Kinesthetic motor imagery training group (Experimental)
  Interventions: Other: Kinesthetic motor imagery training
- Balance exercises (Control) group (Active Comparator)
  Interventions: Other: Balance exercises

INTERVENTIONS:
Other: Dual task training — In addition to balance exercises, random name-word generation, counting the days of the week forward and backward, counting the months of the year forward and backward, subtracting 3 by 3 numbers from 300 to 900 starting from a random number, adding 7 from 1 to 100 and adding 100 Cognitive tasks such as counting tasks by subtracting 7 will be given. While testing dual-task performance, subjects will be asked to perform both tasks without prioritizing and do their best, and will be warned not to stop thinking. In dual-task training, the additional task to be assigned to the motor task will initially be of low complexity and novelty, and will progress to a high degree of complexity and novelty in the training process.
  Arms: Dual task training (balance exercises combined with cognitive task) group
Other: Kinesthetic motor imagery training — Kinesthetic motor imagery training will be planned according to the PETTLEP model. In our study, a single standard motor imagery frame will be created for the subjects. Before starting the motor imagery sessions, individuals will be given an introductory motor imagery session. How to visualize from first-person and third-person perspectives will be explained practically. Motor imagery training will be done in a quiet environment with the door and window closed in order to minimize the external factors that will distract the individual and prevent him from focusing, and the individual will be asked to sit in the motor imagery training sessions. a comfortable chair in the position they feel most comfortable in. Individuals will have their eyes closed throughout the entire motor imagery training. At the beginning of the session, approximately 5 minutes of relaxation exercise will be performed to maximize attention during motor imagery.
  Arms: Kinesthetic motor imagery training group
Other: Balance exercises — Balance exercises will begin with approximately 5 minutes of warm-up exercises and will end with approximately 5 minutes of cool-down exercises at the end of each session. Balance exercises; Static standing on flat ground for 30 seconds with feet together, standing in tandem position for 30 seconds, standing on one leg for 30 seconds, and toes for 30 seconds, one foot airborne backwards, one foot airborne knee flexion slightly squat, one foot airborne knee extension slightly squat, going on the toes, turning with the heel, and multi-directional stretching exercises with eyes open and closed on one leg on the balance board. Each exercise will be performed with 10 repetitions for both lower extremities. Exercises will be applied once a day, 3 days a week for 6 weeks. The exercise program will be accompanied by a physiotherapist and groups of 6-10 people with similar suitability will be formed for the session hours.
  Arms: Balance exercises (Control) group

SUMMARY:
The goal of this clinical trial is to investigate the effects of kinesthetic motor imagery training and dual-task training on cognitive and motor functions in healthy young people. The main question[s] it aims to answer are:

* Kinesthetic motor imagery training and dual-task training do not affect cognitive and motor functions in healthy young people.
* Kinesthetic motor imagery training and dual-task training affect cognitive and motor functions in healthy youth.
* In healthy young people, kinesthetic motor imagery training is more effective on cognitive functions than dual-task training.
* In healthy young people, dual task training is more effective on motor functions than kinesthetic motor imagery training.

Participants will be divided into 3 groups, taking into account the inclusion and exclusion criteria. Participants in each group will be asked to fill out the sociodemographic form before starting the training. Then, initial assessments were the Motion Image Questionnaire-3 to measure motor imagery ability, and the Box and Block Test for mental stopwatch; Stroop Test to measure cognitive functions; In order to evaluate the dual-task performance, the measurement of the dual-task effect and the Berg Balance scale, which evaluates balance as a motor function, and the Y test, which is frequently used in healthy individuals, will be applied. In the balance exercises group, the participants will do the determined balance exercises 3 days a week for 6 weeks, accompanied by a physiotherapist. In the double-task training group, the participants will perform the cognitive tasks in addition to the determined balance exercises, 3 days a week for 6 weeks, accompanied by a physiotherapist. In kinesthetic motor imagery group, the participants will do the physically determined balance exercises in the first session. Participants will participate in imagery exercises, 3 sessions a week for 6 weeks. Visualization studies will be performed in a quiet environment with the eyes closed, accompanied by a physiotherapist, and whether the participants perform a real motor imagery will be examined by evaluating their autonomic functions. At the end of 6 weeks, initial evaluations will be repeated in all groups.

The investigators will compare dual-task training group, kinesthetic motor imagery training group and balance exercises group to see if changes in cognitive and motor function.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18 and 25,
* Absence of a known disease (neurological, mental, orthopedic, vestibular, visual, systemic),
* Unfamiliar with the evaluation and use of motor imagery,
* Individuals who agree to the objectives of this study and to participate voluntarily.

Exclusion Criteria:

* Those who have taken oral corticosteroids or antibiotics within a month,
* Presence of diagnosed systemic or neurological disease.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Information Form | a day before the rehabilitation
  The sociodemographic information of the healthy individuals included in the study will be obtained first with the form prepared by us. Questionnaire; It will contain information about the individual's age, gender, weight, height, educational status, occupation, socioeconomic status, employment status, marital status, drug use, psychological disorders and chronic diseases of the individual.
Motion Imagery Questionnaire-3 | a day before the rehabilitation
  The Motion Imagination Questionnaire-3, The Motion Imagination Questionnaire, and the Motion Imagination Questionnaire- Revised, 2nd Edition is the most current version. In the questionnaire consisting of 12 items, external, internal and kinesthetic visualization abilities are evaluated separately. The Turkish validity and reliability of the questionnaire was determined by Dilek et al. made by It consists of 3 subscales and a total of 12 items evaluating external visual imagery, internal visual imagery and kinesthetic imagery. Each of the 12 tasks in the questionnaire will be performed physically first, then the participant will return to the starting position and imagery will be performed according to the desired imagery type. The scoring will be between 1 and 7, with 1 point: very difficult to see/feel, 7 points: very easy to see/feel.
Motion Imagery Questionnaire-3 | after 6 weeks of training
  The Motion Imagination Questionnaire-3, The Motion Imagination Questionnaire, and the Motion Imagination Questionnaire- Revised, 2nd Edition is the most current version. In the questionnaire consisting of 12 items, external, internal and kinesthetic visualization abilities are evaluated separately. The Turkish validity and reliability of the questionnaire was determined by Dilek et al. made by It consists of 3 subscales and a total of 12 items evaluating external visual imagery, internal visual imagery and kinesthetic imagery. Each of the 12 tasks in the questionnaire will be performed physically first, then the participant will return to the starting position and imagery will be performed according to the desired imagery type. The scoring will be between 1 and 7, with 1 point: very difficult to see/feel, 7 points: very easy to see/feel.
Box and Block Test (Mental Stopwatch Measurement) | a day before the rehabilitation
  Box and Block Test is a test developed to measure rough manual dexterity. The equipment used in the study was divided into two 25.4 cm sections with a 15.2 cm high divider in accordance with the adult norms previously determined in the literature. In the study, unlike the original procedure of the test, it is not the number of blocks collected in a limited time; The time required to collect 15 blocks will be recorded. The purpose of this change; In this study, it is aimed to evaluate mental chronometry ability rather than manual skill. Individuals will first be asked to physically move 15 blocks to the other section, and the elapsed time will be recorded. The application will be made with the dominant party. After the materials are removed from the field of view of the individuals, they will be asked to perform this transport activity with the imaging method and to report when they place each block during imaging and the elapsed time will be recorded .
Box and Block Test (Mental Stopwatch Measurement) | after 6 weeks of training
  Box and Block Test is a test developed to measure rough manual dexterity. The equipment used in the study was divided into two 25.4 cm sections with a 15.2 cm high divider in accordance with the adult norms previously determined in the literature. In the study, unlike the original procedure of the test, it is not the number of blocks collected in a limited time; The time required to collect 15 blocks will be recorded. The purpose of this change; In this study, it is aimed to evaluate mental chronometry ability rather than manual skill. Individuals will first be asked to physically move 15 blocks to the other section, and the elapsed time will be recorded. The application will be made with the dominant party. After the materials are removed from the field of view of the individuals, they will be asked to perform this transport activity with the imaging method and to report when they place each block during imaging and the elapsed time will be recorded .
Stroop Test | a day before the rehabilitation
  It is a test that evaluates frontal lobe functions and cognitive processes such as attention, information processing, and resistance to interference. In the application consisted of 5 sections. The times obtained by the participants in each section will be noted in the section on the registration form. For incorrect responses by the participants, a slash (/) will be drawn over the relevant letter in the registration form; When participants correct their mistakes on their own, the relevant items will be circled (O). The performance of the participants will be scored according to three separate criteria for each section: (1) the time taken until the "start" command and the last item of the section are answered; (2) the number of errors; (3) the number of corrected responses. The minimum time to complete the reading/saying process for each section, the "0" error score and the "0" number of corrections determine the highest score that can be obtained from the Stroop Test.
Stroop Test | after 6 weeks of training
  It is a test that evaluates frontal lobe functions and cognitive processes such as attention, information processing, and resistance to interference. In the application consisted of 5 sections. The times obtained by the participants in each section will be noted in the section on the registration form. For incorrect responses by the participants, a slash (/) will be drawn over the relevant letter in the registration form; When participants correct their mistakes on their own, the relevant items will be circled (O). The performance of the participants will be scored according to three separate criteria for each section: (1) the time taken until the "start" command and the last item of the section are answered; (2) the number of errors; (3) the number of corrected responses. The minimum time to complete the reading/saying process for each section, the "0" error score and the "0" number of corrections determine the highest score that can be obtained from the Stroop Test.
Evaluation of Dual- Task Performance | a day before the rehabilitation
  In order for dual-task performance to be fully evaluated, both tasks must be evaluated separately and then as a dual-task before and after rehabilitation. The tasks given in our study will be evaluated one by one before the application. In our study, dual-task performance will be measured by calculating the 'dual-task effect' for both tasks.
  If the result is positive, there is an improvement in dual-task conditions; negative, it will be considered a reduction in dual-task conditions. Positive dual-task effect values show the relative improvement in dual-task performance; negative dual-task effect values indicate worsening of performance in dual-task compared to single-task.
Evaluation of Dual- Task Performance | after 6 weeks of training
  In order for dual-task performance to be fully evaluated, both tasks must be evaluated separately and then as a dual-task before and after rehabilitation. The tasks given in our study will be evaluated one by one before the application. In our study, dual-task performance will be measured by calculating the 'dual-task effect' for both tasks.
  If the result is positive, there is an improvement in dual-task conditions; negative, it will be considered a reduction in dual-task conditions. Positive dual-task effect values show the relative improvement in dual-task performance; negative dual-task effect values indicate worsening of performance in dual-task compared to single-task.
Y Balance Test | a day before the rehabilitation
  Star Shaped Sudden Change Balance Test is a test that measures balance dynamically that requires strength, flexibility and proprioception. Y Balance test is a modified version of this test. This modified test includes extensions in the anterior, posteromedial, and posterolateral directions. The test procedures will be set up on a flat surface with 3 measuring tapes so that the angle between the posteromedial-posterolateral direction is 90˚ and the angle between the anterior and posterior directions is 135˚. The individual will be asked to stand on one foot at the midpoint of the test setup and touch the anterior, posteromedial and posterolateral directions with the other foot while maintaining the correct balance with the tip of the toe. The test will be repeated 3 times in all directions, averaged and recorded in cm. The score will be obtained by taking the average of 3 elongation for each direction, dividing this average by the leg length and multiplying by 100.
Y Balance Test | after 6 weeks of training
  Star Shaped Sudden Change Balance Test is a test that measures balance dynamically that requires strength, flexibility and proprioception. Y Balance test is a modified version of this test. This modified test includes extensions in the anterior, posteromedial, and posterolateral directions. The test procedures will be set up on a flat surface with 3 measuring tapes so that the angle between the posteromedial-posterolateral direction is 90˚ and the angle between the anterior and posterior directions is 135˚. The individual will be asked to stand on one foot at the midpoint of the test setup and touch the anterior, posteromedial and posterolateral directions with the other foot while maintaining the correct balance with the tip of the toe. The test will be repeated 3 times in all directions, averaged and recorded in cm. The score will be obtained by taking the average of 3 elongation for each direction, dividing this average by the leg length and multiplying by 100.
Berg Balance Scale | a day before the rehabilitation
  Berg balance scale is a frequently used and easily applicable scale to evaluate static and dynamic balance in adults, consisting of fourteen instructions. The highest possible score is 56 points. 0-20 points indicate balance disorder, 21-40 points indicate an acceptable balance, and 41-56 points indicate a good balance. It takes about 10 to 20 minutes to complete the scale.
Berg Balance Scale | after 6 weeks of training
  Berg balance scale is a frequently used and easily applicable scale to evaluate static and dynamic balance in adults, consisting of fourteen instructions. The highest possible score is 56 points. 0-20 points indicate balance disorder, 21-40 points indicate an acceptable balance, and 41-56 points indicate a good balance. It takes about 10 to 20 minutes to complete the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, Centre, Turkey (Türkiye)

REFERENCES:
- [Background] Sarasso E, Agosta F, Piramide N, Gardoni A, Canu E, Leocadi M, Castelnovo V, Basaia S, Tettamanti A, Volonte MA, Filippi M. Action Observation and Motor Imagery Improve Dual Task in Parkinson's Disease: A Clinical/fMRI Study. Mov Disord. 2021 Nov;36(11):2569-2582. doi: 10.1002/mds.28717. Epub 2021 Jul 19. PMID 34286884
- [Result] Mencel J, Marusiak J, Jaskolska A, Kaminski L, Kurzynski M, Wolczowski A, Jaskolski A, Kisiel-Sajewicz K. Motor imagery training of goal-directed reaching in relation to imagery of reaching and grasping in healthy people. Sci Rep. 2022 Nov 3;12(1):18610. doi: 10.1038/s41598-022-21890-1. PMID 36329083
- [Result] Kahraman T, Kaya DO, Isik T, Gultekin SC, Seebacher B. Feasibility of motor imagery and effects of activating and relaxing practice on autonomic functions in healthy young adults: A randomised, controlled, assessor-blinded, pilot trial. PLoS One. 2021 Jul 13;16(7):e0254666. doi: 10.1371/journal.pone.0254666. eCollection 2021. PMID 34255812